CLINICAL TRIAL: NCT03460951
Title: MRI of the Brachial Plexus and Chronic Inflammatory Demyelinating Polyradiculoneuropathy: Assessment of DTI-derived Measurements at 3.0-T
Brief Title: Diffusion Tensor Imaging in Chronic Inflammatory Demyelinating Polyneuropathy (PIDC)
Acronym: PIDC
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-379; 2013-A00808-37 (Other: 2013-A00808-37)
Record Dates: First submitted 2018-02-16; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: CIDP (Chronic Inflammatory Demyelinating Polyradiculoneuropathy); CMT (Charcot Marie Tooth Disease)
Keywords: Feasibility and reproductibility; DTI parameters (Fractional Anisotropy, Apparent Diffusion Coefficient); MRI morphological parameters (T1, STIR)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CIDP patients: 15 patients with CIDP (Chronic Inflammatory Demyelinating Polyradiculoneuropathy ) who satisfy the definite CIDP criteria of the Joint Task Force of the EFNS and PNS 1 (situations A and B according to the French CIDP work group2), and who agree to undergo cervical MRI.
  Interventions: Diagnostic Test: cervical MRI
- Normal volunteers: 15 healthy subjects matched for age and gender to CIDP patients
  Interventions: Diagnostic Test: cervical MRI
- Charcot-Marie-Tooth disease type 1A patients (CMT-1A): 15 CMT-1A patients (proven by genetic testing), will be included as Charcot-Marie-Tooth disease type 1A patients (CMT-1A) is one of the main differential diagnoses of CIDP characterized by the diffuse demyelination of peripheral nerves.
  Interventions: Diagnostic Test: cervical MRI

INTERVENTIONS:
Diagnostic Test: cervical MRI — Cervical MRI will be performed in all of the patients and controls on a 3.0-T scanner (Discovery MR750, General Electric (GE) Medical Systems, Milwaukee, WI, USA)

SUMMARY:
The main purpose of this study is to assess the clinical feasibility of diffusion tensor imaging (DTI) for the diagnosis of chronic inflammatory demyelinating polyradiculoneuropathy (CIDP). For thar purpose, investigator will compare, fractional anisotropy (FA) obtained by diffusion tensor imaging (DTI) MRI 3T on brachial plexus and cervical spinal nerve roots between patients with defined Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), according to the EFNS 2010 criteria, and healthy controls.

The secondary outcomes will be to compare DTI parameters (FA, ADC or Apparent Diffusion Coefficient) between CIDP patients, healthy volunteers, and patients with Charcot Marie Tooth disease type 1a (CMT1a) and MRI morphological parameters (T1, STIR) between these groups. Moreover, investigator will investigate the possible relationship between MRI parameters, clinical indices, and electrophysiological measure.

DETAILED DESCRIPTION:
Investigator will prospectively enroll 15 patients with CIDP followed in the Neurology Department of Clermont Ferrand University Hospital, who satisfy the Joint Task Force of the EFNS and PNS definite CIDP criteria. Two control groups will be studied in parallel, including 15 healthy volunteers on one side, and 15 patients with CMT-1A on the other side (proven by genetic testing). Using a 3-T magnetic resonance imaging scanner, we will obtain DTI scans of brachial plexus of these 3 groups, prepare fractional anisotropy (FA) maps, and compare these values between groups. Investigator will evaluate MRI imaging findings too (coronal STIR, T1-weighted images,and DWIs). MRI studies will be reviewed independently by two neuroradiologists, blinded to clinical informations. In all patients with CIDP, investigator will also performs clinical evaluation and electroneuromyography. Correlation between FA values clinical indices will be examined.

ELIGIBILITY:
Inclusion Criteria:

* - For All patients: at least 18 years-old.
* For CMT1a group : CMT1 a should be proven by genetic testing
* For CIDP group: CIDP should satisfied the definite CIDP criteria of the Joint Task Force of the EFNS and PNS 1 (situations A and B according to the French CIDP work group2). They might have received steroids, immunoglobulin or immunosuppressive treatments

Exclusion Criteria:

* For all groups: any neurological comorbidity, other causes of neuropathy or history of exposure to neurotoxic agents (the inclusion and exclusion criteria are detailed in supplemental data) allergies, renal failure, Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men or women
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Fractional Anisotropy in C5 to C8 nerve roots in CIDP patients compared to CMT-1A patients and healthy controls. | At day 1
  Diffusion Tensor Imaging (DTI) is a modality of Diffusion-Weighted Imaging (DWI). Fractional Anisotropy (FA) and Apparent Diffusion Coefficient (ADC) values, determines the magnitude of directionality of diffusion.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficient (ADC) values in C5 to C8 nerve roots in CIDP patients compared to CMT-1A patients and healthy controls | At day 1
  Diffusion Tensor Imaging (DTI) is a modality of Diffusion-Weighted Imaging (DWI). Fractional Anisotropy (FA) and Apparent Diffusion Coefficient (ADC) values, determines the magnitude of directionality of diffusion.
Cervical nerve roots diameter | at day 1
  The diameters of cervical nerve roots (C6-C8) will be measured at the outlet of the intervertebral canal, on coronal STIR sequences, using an ADW 4.5 workstation.
Clinical data analysis | at day 1
  Disease severity at inclusion (Medical Research Council score (MRC), INCAT sensory sum score (INCAT), Overall Neuropathy Limitation Scale (ONLS)) will be prospectively assessed by the same study investigator. We will also perform nerve conduction studies on all the CIDP patients
Electrophysiological data analysis : motor conduction | at day 1
  Amplitude of compound muscle action potential (ACMAP),
Electrophysiological data analysis motor conduction | at day 1
  Motor conduction velocity (MCV)
Electrophysiological data analysis motor conduction | at day 1
  Motor distal latency (MDL)
Electrophysiological data analysis motor conduction | at day 1
  F-wave latency (FL)
Electrophysiological data analysis :motor conduction | at day 1
  terminal latency index (TLI))
Electrophysiological data analysis : sensitive conduction | at day 1
  Amplitude of sensitive potential (ASP)
Electrophysiological data analysis : sensitive conduction | at day 1
  Sensitive conduction velocity (SCV)
Electrophysiological data analysis : sensitive conduction | at day 1
  Sensitive distal latency (SDL)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric TAITHE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France